CLINICAL TRIAL: NCT00001204
Title: Cardiovascular Evaluation of Homozygous Familial Hypercholesterolemia
Brief Title: Cardiovascular Evaluation of Patients With High Cholesterol and Normal Volunteers
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 850105; 85-H-0105
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-08-19

CONDITIONS: Homozygous Familial Hypercholesterolemic
Keywords: Dyslipoproteinemia; Hypercholesterolemia; Atherosclerosis; Natural History
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Longitudinal sequential cardiologic studies utilizing noninvasive techniques in homozygous patients with well-characterized LDL receptor defects

SUMMARY:
Homozygous familial hypercholesterolemia is a rare inherited disease of metabolism. It occurs in less than 1 in 1 million people within the United States. Patients with the disease are typically children and young adults who develop heart disease early in life. Children less than age 5 years with this disease have suffered heart attacks and death.

The normal process that removes cholesterol particles from the blood stream does not work in patients with this disease. It causes cholesterol to build-up in the arteries and leads to hardening of the arteries (atherosclerosis).

The goal of this study is to detect and measure atherosclerosis in these patients before it becomes permanent and potentially life threatening. Patients with this disease can participate in this study. Researchers plan to evaluate patients with homozygous familial hypercholesterolemia using new and standard methods for detecting atherosclerosis.

Researchers plan to use information gathered during this study to develop new, promising treatments such as liver transplantation and gene therapy.

DETAILED DESCRIPTION:
Familial hypercholesterolemia is an autosomal co-dominant disorder resulting in abnormal LDL receptor function, profoundly elevated concentrations of low density lipoproteins, accelerated atherosclerosis and death by early adulthood. This disease is heterogeneous in both the degree of LDL receptor dysfunction as well as the age of death. Liver transplantation has been demonstrated to virtually normalize plasma lipoprotein concentrations in homozygous FH and the recent cloning of a functional LDL receptor gene holds promise in the definitive treatment of this condition. We propose performing longitudinal sequential cardiologic studies utilizing noninvasive techniques in homozygous patients with well-characterized LDL receptor defects. Sequential cardiovascular study of these patients will not only characterize the progression of atherosclerosis heart disease in this disease, it may also permit the identification of individuals with would be likely to benefit from liver transplantation and/or genetic engineering.

ELIGIBILITY:
* INCLUSION CRITERIA:

Fasting cholesterol greater than 500 mg/dl, low density lipoprotein cholesterol greater than 400 mg/dl, and triglycerides less than mg/dl.

Family history of hypercholesterolemia and/or cardiovascular disease before the age of 60 years.

Tendinous and tuberous xanthomas.

Arcus corneae before the age of 30.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Familial hypercholesterolemia
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 1992-01-07 (Actual)

PRIMARY OUTCOMES:
We propose performing longitudinal sequential cardiologic studies utilizing noninvasive techniques in homozygous patients with well-characterized LDL receptor defects. | one year
  Descriptive data

SECONDARY OUTCOMES:
Current work has focused on identifying new noninvasive measurements of CAD and quantitating atherosclerosis burden. | one year
  Current work has focused on identifying new noninvasive measurements of CAD and quantitating atherosclerosis burden.

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Shamburek, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hoeg JM. Familial hypercholesterolemia. What the zebra can teach us about the horse. JAMA. 1994 Feb 16;271(7):543-6. doi: 10.1001/jama.271.7.543. No abstract available. PMID 8301770
- [Background] Sprecher DL, Hoeg JM, Schaefer EJ, Zech LA, Gregg RE, Lakatos E, Brewer HB Jr. The association of LDL receptor activity, LDL cholesterol level, and clinical course in homozygous familial hypercholesterolemia. Metabolism. 1985 Mar;34(3):294-9. doi: 10.1016/0026-0495(85)90015-0. PMID 3856094
- [Background] Schmidt HH, Hill S, Makariou EV, Feuerstein IM, Dugi KA, Hoeg JM. Relation of cholesterol-year score to severity of calcific atherosclerosis and tissue deposition in homozygous familial hypercholesterolemia. Am J Cardiol. 1996 Mar 15;77(8):575-80. doi: 10.1016/s0002-9149(97)89309-5. PMID 8610605
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1985-H-0105.html